CLINICAL TRIAL: NCT03503994
Title: A Dose-Ranging Study to Assess the Effect of Inhaled Corticosteroids in Ventilated Preterm Neonates
Brief Title: Inhaled Corticosteroids for Treatment of Bronchopulmonary Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); IWK Health Centre (Other)
Responsible Party: Principal Investigator, Vibhuti Shah, Staff Neonatologist, Mount Sinai Hospital, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000/363
Record Dates: First submitted 2018-03-30; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drug (Other): Patients receiving inhaled beclomethasone diproprionate in four escalating doses:
  1. 200 mcg bid
  2. 400 mcg bid
  3. 600 mcg bid
  4. 800 mcg bid
  Interventions: Drug: Inhaled Beclomethasone Dipropionate Monohydrate

INTERVENTIONS:
Drug: Inhaled Beclomethasone Dipropionate Monohydrate — Beclomethasone Dipropionate (HFA-BDP, QVAR*) in the following doses will be evaluated:
  1. 200 mcg bid
  2. 400 mcg bid
  3. 600 mcg bid
  4. 800 mcg bid

SUMMARY:
While many short-term morbidities associated with extreme prematurity have declined over the last two decades, the incidence of bronchopulmonary dysplasia (BPD) has increased to a rate of approximately 45% in neonates <28 weeks gestational age (GA) and birth weight (BW) <1,500 g. Neonates with BPD are at increased risk for adverse short-and long-term neurodevelopmental and respiratory outcomes that often persist into adulthood.

There is a growing body of pathological and biochemical evidence that implicates inflammation in its pathogenesis. This is further supported by randomized controlled trials (RCTs) that demonstrate the efficacy of systemic corticosteroids in facilitating extubation and reducing BPD. However, several short- and long-term adverse effects associated with the use of systemic corticosteroids have been described, the most concerning of which is their effect on neurodevelopment, specifically an increased rate of cerebral palsy (CP).

Inhaled corticosteroids (ICS) are an attractive alternative to systemic steroids because of these concerns. Earlier systematic reviews had not found any benefit in using ICS for the prevention or treatment of BPD. However, a recent systematic review showed a significant reduction in death or BPD at 36 weeks' corrected GA (CGA) (risk ratio=0.86, 95% confidence interval 0.75, 0.99), BPD (RR=0.77, 95% CI 0.65, 0.91), and use of systemic steroids (RR=0.87, 95% CI 0.76, 0.98) in infants treated with ICS.

Despite growing evidence of the effectiveness of ICS for BPD, uncertainty remains over treatment timing, effective dose, and long-term effects. There is also variation in the delivery systems used for delivery of ICS. These concerns continue to be echoed in a recent review by Nelin et al. Given that the long-term neurodevelopmental impact of ICS were unknown at the time of this study and many infants are able to wean from ventilation without steroids, the investigators conducted an escalating-dose ranging study of late ICS (i.e. administered after the first week of life) delivered by a metered dose inhaler (MDI) utilizing a specially designed valved delivery system to determine the minimum effective dose necessary to achieve extubation or reduction in oxygen requirements and the long-term neurodevelopmental impact of increasing doses of ICS.

DETAILED DESCRIPTION:
Research Question:

What is the effective dose of inhaled steroids (HFA-BDP) in ventilated preterm infants? Material and Methods Objective: The primary purpose of this study is to determine the optimal dose of inhaled steroids (using HFA-BDP) in ventilated preterm infants. The result from this study will determine the dose of inhaled steroids to be used for a subsequent randomized placebo-controlled trial with sufficient power to determine if inhaled steroid is associated with reduction in CLD in ventilated preterm infants without any detrimental effect on long term neurodevelopmental outcome.

Study Design: Escalating dose-ranging study Study Population: Babies with birth weights < 1,250 grams and gestational age < 32 weeks admitted in the NICU at Sunnybrook and Women's College Health Sciences Centre and Mount Sinai Hospital Inclusion Criteria: Birth weight < 1,250 grams and gestational age < 32 weeks, Need for assisted mechanical ventilation (ventilation rate > 15 breaths/min, and fractional oxygen concentration of inspired gas (Fio2) > 0.3 but < 0.6), Postnatal age 10-21 days, Stable ventilatory requirements over the 48-72 hours prior to enrollment Exclusion Criteria: Actual or suspected sepsis, Congenital cardiorespiratory malformation, Patent ductus arteriosus, Presence of necrotizing enterocolitis, gastrointestinal hemorrhage or perforation, Treatment with systemic dexamethasone Duration of therapy: 7 days Drug Regimen: Groups of neonates will be treated with an escalating dose of HFA-BDP until either efficacy equal to that seen with dexamethasone or significant side-effects are observed. 10 neonates will be treated at each dosage level before moving up to the next dose. Each neonate will be treated with only one dose.

Bowser et al have performed an in vitro evaluation of drug deposition of HFA-BDP (QVAR*) and CPC-BDP MDI (Beclovent) via an aerosol delivery chamber (Aerochamber) and endotracheal tube (uncuffed Portex 3.5, 3.0 and 2.5) at low tidal volumes. The PARI Compas Breath Simulator was used to simulate neonatal and infant respiratory cycles. For both formulations and all endotracheal tubes, the output (*g) increased significantly at the tidal volume and inspiratory flow rates were increased. The 3.5 endotracheal tube side gave greater output/puff at all tidal volumes and for both formulations as compared to the smaller endotracheal tubes. Greater in vitro deposition was measured for QVAR than for beclovent, possibly leading to greater in vivo delivery to the lung of this new HFA-BDP MDI formulation to intubated infants

Thus, for the purpose of this study Beclomethasone Dipropionate (HFA-BDP, QVAR*) in the following doses will be evaluated:

1. 200 *g bid
2. 400 *g bid
3. 600 *g bid
4. 800 *g bid Inhaled steroids will be administered using a specially designed neonatal aerosol delivery system manufactured by Trudell Canada (see diagram, Appendix I). The device will be connected directly to the endotracheal tube on one side with the ventilator circuit on the other. The ventilator settings will be temporarily adjusted to achieve an expiratory tidal volume of 7ml/kg (based on birth weight) and a rate of 30 breaths/min and an inspiratory time of 0.5 seconds. There will be a one-minute interval between each actuation from the MDI. Continuous cardiac and oxygen saturation monitoring will be used throughout the treatment period. One-minute after the final puff has been administered, the delivery system will be removed and the baby returned to the ventilator settings previously used. The total daily dose will be administered in two divided doses.

If the infant is extubated during the study period administration of inhaled medications will be stopped.

Outcome Measures - Efficacy Primary Outcome: Reduction in Fio2 from the 2 days prior to treatment to the final 2 days of the study period or extubation during the study period. Extubation is considered to be successful if the infant does not require assisted ventilation in the next 48 hours. A reduction in additional Fio2 of 75% or greater will be considered a significant improvement (i.e. a baby with a baseline Fio2 of 0.51 who requires less than 0.28 [0.21 + 0.25 (0.51-0.21)] at the end of the treatment period will be considered a treatment success).

Secondary Outcome:

Ventilatory status: Ventilator rate Mean airway pressure Peak inspiratory pressure Ventilatory parameters will be assessed at the same time intervals as Fio2 described above.

Adverse Event Monitoring Each patient will be carefully monitored for adverse events by the investigators. The following events will be specifically monitored.

1. Hypertension: Blood pressure (BP) will be noted every 12 hourly using an automatic sphygmomanometer (Dinamap, Criticon Inc.). Hypertension is defined as BP higher than 2 SD above the mean for the infant's gestational and postnatal age.
2. Hyperglycemia: Urine and blood glucose will be monitored as per nursing standard protocol for infants who are on steroids. Hyperglycemia will be defined as a blood glucose > 10 *mol/L.
3. Growth: Weight and head circumference will be recorded prior to and after completion of the study period.
4. Infection: Sepsis is defined as a need for antibiotic therapy because of a positive blood or cerebrospinal fluid culture or clinical diagnosis of pneumonia.
5. Evidence of feeding intolerance, necrotizing enterocolitis or intestinal perforation will be noted.
6. Candidiasis of the mouth and throat will be noted. Assessment will be made of the seriousness, intensity and relationship to the administration of the study medication. If, in the opinion of the investigator, the adverse event is not tolerated, the patient will be withdrawn from the study and monitored until resolution of the adverse event or until a conclusion is reached as to its irreversible nature.

Suppression of the hypothalamic-pituitary-adrenal axis (HPA):

Adrenal suppression is an important adverse effect, which occurs during glucocorticoid therapy (particularly when administered systemically). Controversy exists regarding the variable effect of glucocorticoid therapy on the immature HPA axis. The dose and duration of therapy, methodology and timing of adrenal function assessment and inter-patient variablity influence the degree and duration of suppression. Also, there is no consensus regarding normal HPA function in extremely premature infant. Therefore, for the purpose of this pilot study where the drug is administered for a very short duration the HPA axis will not be investigated. Assessment of the HPA axis will be part of the larger randomized controlled trial.

Laboratory test abnormalities considered by the Investigator to be clinically relevant will be reported on the Adverse Event Page of the CRF.

Adverse events and laboratory test abnormalities fulfilling the definition of "serious" must, in addition, be reported in detail on the Serious Adverse Event Form.

Signs and symptoms of each AE should be described in detail: start and stop dates, intensity, relationship it investigational product, action taken and outcome.

Safety Assessment Adverse events will be tracked as described below. After each serious AE, the safety monitoring committee will be informed and will investigate the relationship between the AE and study drug administration. Any time a serious AE is felt to be "probably related" to the therapy, consideration will be given to stopping the study. If a series of serious AE events are felt to be "possibly related" or a series of minor events felt to be "probably related" to treatment with the study drug, the study may also be stopped. The REB, 3M pharmaceuticals and HPB will be kept informed of all such deliberations. The members of the safety committee include Dr. Arne Ohlsson, Director Evidence Based Neonatal Care and Outcomes Research, MSH, Dr. Elizabeth Asztalos, Staff Neonatologist, SWCHSC and Joseph Beyene, Biostatistician, MSH. After enrollment of 10 neonates at a particular dosing level the safety committee will be requested to review the data for efficacy and safety. If no benefit or no significant adverse events are noted then the decision will be made to move to the next dosing level.

Weaning Protocol Respiratory therapists will use set criteria for weaning from ventilation. For 48 hours prior to commencement of treatment, a record will be made of the baseline ventilator settings. A transcutaneous pCO2 monitor will be applied daily for the duration of the study. Blood gases (capillary or arterial) will be performed as clinically indicated: ie. in response to changes in clinical status, oxygen requirements (oxygen saturation) or transcutaneous pCO2. Supplemental oxygen and ventilation will be adjusted to maintain an oxygen saturation of 90-95%, carbon dioxide tension between 45-60mm Hg (5.8-7.8 KPA) and a blood pH of at least 7.25. If clinically indicated, the proximal airway pressure will be reduced in decrements of 2mm Hg until a mean airway pressure of 8mm Hg is reached, following which the ventilator rate will be reduced in decrements of 2-5 breaths/min until a rate of 10-12 breaths/min is achieved. Neonates will be extubated from a rate of 10-12 breaths/min a mean airway pressure of 8mm Hg and Fio2 concentration of < 0.3. A record will be made of the need for nasal CPAP following extubation.

Sample size estimation The study design is an escalating dose ranging study with an aim to identify both an effective and a safe dose of inhaled steroids. 10 babies will be enrolled in each dose category. The study will be stopped if the therapeutic efficacy is achieved in a given dosage group or if significant side effects are noted. Therapeutic efficacy will be considered to have occurred in a group of 6 or more babies out of 10 meet the primary outcome [based upon response expected with dexamethasone therapy - data from Ohlsson et al (Unpublished data from MSc thesis)].

Statistical Analysis Analysis of variance for repeated measures will be used to assess the effect of therapy over time in each dosage group. This analysis will be applied to Fio2 and ventilatory parameters

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 1,250 grams
* Gestational age < 32 weeks
* Need for assisted, invasive mechanical ventilation with at least the following settings:

ventilation rate > 15 breaths per min, fractional oxygen concentration of inspired gas (FiO2) > 30% but < 60%)

* Postnatal age 10-21 days
* Stable ventilatory requirements over the 48-72 hours prior to enrollment

Exclusion Criteria:

* Actual or suspected sepsis
* Congenital cardiorespiratory malformation
* Patent ductus arteriosus
* Presence of necrotizing enterocolitis
* Presence of gastrointestinal hemorrhage or perforation
* Treatment with systemic dexamethasone

Ages: 1 Week to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2001-07-27 (Actual); Primary Completion 2006-11-15 (Actual); Study Completion 2006-11-15 (Actual)

PRIMARY OUTCOMES:
Reduction in FiO2 > 75% | 1 week per dose
  Reduction in FiO2 (%) from the 2 days prior to treatment to the final 2 days of the study period. A reduction in additional FiO2 of 75% or greater will be considered a significant improvement. For example, a baby with a baseline FiO2 of 51% would have a significant reduction in FiO2 if post-treatment FiO2 is less than 0.28 using the following calculation: FiO2 reduction 75% = [0.21 + 0.25 (0.51-0.21)]
Successful extubation | 1 week per dose
  Extubation during the study period is considered to be successful if the infant does not require assisted, invasive ventilation for at least 48 hours after the removal of the endotracheal tube and is extubated during the treatment period.

SECONDARY OUTCOMES:
Ventilator rate (breaths per minute) | 1 week
  Ventilator rate (breaths per minute) at the end of treatment
Mean airway pressure (cm H2O) | 1 week
  The mean airway pressure (cm H2O) required by the baby at the end of treatment
Peak inspiratory pressure (cm H2O) | 1 week
  The peak inspiratory pressure (cm H2O) required by the baby at the end of treatment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raghuram K, Dunn M, Jangaard K, Reilly M, Asztalos E, Kelly E, Vincer M, Shah V. Inhaled corticosteroids in ventilated preterm neonates: a non-randomized dose-ranging study. BMC Pediatr. 2018 May 7;18(1):153. doi: 10.1186/s12887-018-1134-7. PMID 29734948